CLINICAL TRIAL: NCT04082884
Title: Very Low Carbohydrate Diet as an Adjunctive Therapy for Youth Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2000026189; 2K12DK094714-06 (NIH)
Record Dates: First submitted 2019-09-06; First posted 2019-09-09 (Actual); Results first posted 2023-06-05 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Type 1 Diabetes
Keywords: very low carbohydrate diet
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Following enrollment, participants will follow a standard carbohydrate diet for 2 weeks. They will then undergo a 1 week transition followed by 2 weeks on a higher protein very low carbohydrate diet that is then followed by 2 weeks on a higher fat very low carbohydrate diet.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Very Low Carbohydrate Diet (Experimental): Participants will follow a high protein very low carbohydrate diet (VLCD) for 2 weeks. This will be 11% of caloric intake from carbohydrates, 54% of calories from protein, and 35% of calories from fat. Immediately following this, participants will follow a high protein very low carbohydrate diet (VLCD) which will be 11% of caloric intake from carbohydrates, 23% of calories from protein, and 66% of calories from fat.
  Interventions: Behavioral: Very Low Carbohydrate Diet

INTERVENTIONS:
Behavioral: Very Low Carbohydrate Diet — A very low carbohydrate diet (VLCD), is defined as limiting carbohydrate intake to 11% of total daily caloric intake.

SUMMARY:
This prospective, open-label pilot/feasibility study of 10 youth with T1D is to evaluate glycemic and metabolic changes taking place with a very low carbohydrate diet.

DETAILED DESCRIPTION:
First, to evaluate the feasibility of following each type of VLCD (high protein or high fat), participants will follow a standard carbohydrate diet for 2 weeks, followed by a 1 week transition to a VLCD, and then follow the a high protein VLCD for 2 weeks followed by a high fat VLCD for 2 weeks. The study will consist of 4 in person or virtual visits which will take place over ~7 weeks. All participants will be initially studied for 2 weeks while ingesting a standard diet recommended by the American Diabetes Association, followed by a 1-week transition to a VLCD, and followed by 2 weeks on each type of VLCD (high protein, high fat). During the first (baseline) period fasting β-hydroxybutyrate levels will be measured 2-3 times per week. During the VLCD study periods, fasting β-hydroxybutyrate levels will be measured daily in the morning using a blood ketone meter; insulin doses will be collected using insulin pump downloads and continuous glucose monitoring (CGM) profiles will be used to assess glycemic excursions on each diet, as well as the time in hypo-, eu- and hyperglycemic ranges. The purpose of this study is to examine changes in sensor glucose levels, basal and bolus insulin doses, and metabolic factors following implementation of a very low carbohydrate diet (VLCD). Sensor-derived time glucose ranges will serve as a surrogate marker of hemoglobin A1c given the short duration of the study. Safety measures of the diet will also be assessed, including daily fasting ketone levels.

The first hypothesis of the study is that use of a VLCD with strict monitoring of ketosis will reduce glycemic variability and increase time in target range, defined as 70-180 mg/dL by reducing the time in the hyperglycemic (>180 mg/dL) and hypoglycemic ranges (<70 mg/dL). Decreased carbohydrate intake will lead to less postprandial hyperglycemia. Lower insulin doses for meals and snacks as a result of decreased carbohydrate intake will lessen postprandial hypoglycemia as well.

ELIGIBILITY:
Inclusion Criteria:

* BMI 19-30 m2 for individuals at least 18 years old or BMI < 95 percentile for individuals less than 18 years old
* Participants 18 years of age must be able to read and provide written consent
* Participants under 18 years of age must be able to read and provide written assent
* Participants are managed using an insulin pump or injections
* Participant has or is willing to wear a CGM for the duration of the study
* Participant is willing to complete diet logging procedures stated above

Exclusion Criteria:

* A1c < 6.5% or > 10%
* Recent history of more than 1 of diabetic ketoacidosis (DKA) in the past 6 months
* Treatment with glucose-lowering drugs other than insulin
* Unstable psychiatric disorders, including eating disorders (DSM-V criteria)
* Weight loss medications within the last 6 months
* Females who are pregnant, lactating or planning to become pregnant in the next 6 months
* Another medical condition that precludes participation in the study

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-02-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Yale-New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Participants: Participants will follow a high protein very low carbohydrate diet (VLCD) for 2 weeks. This will be 11% of caloric intake from carbohydrates, 54% of calories from protein, and 35% of calories from fat. Immediately following this, participants will follow a high fat very low carbohydrate diet (VLCD) which will be with 11% caloric intake from carbohydrates, 23% from protein, 66% from fat.
  Very Low Carbohydrate Diet: A very low carbohydrate diet (VLCD), is defined as limiting carbohydrate intake to 11% of total daily caloric intake.
  The high fat very low carbohydrate diet was removed from the study after the 4th participant completed the study.
Period: Overall Study
Arm/Group | Overall Participants
Started | 6
Completed Standard Diet | 5
1 Week Transition to Low Carbohydrate Diet Completed | 5
High Protein Low Carbohydrate Completed | 5
High Fat Low Carbohydrate Completed | 4
Completed | 5
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall Participants: Participants were youth ages 14-23 with a diagnosis of type 1 diabetes.
Arm/Group | Overall Participants
Number analyzed (Participants) | 6
Age, Customized [Count of Participants; unit: Participants]
  Age in years categorized: 10-19 years | 3
  Age in years categorized: 20-29 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time in Target Range of 70-180 mg/dL.
Description: The target range is 70 mg/dL - 180 mg/dL based on sensor-derived glucose levels. The outcome is reflected as the percentage of time spent in this range during the time frame.
Time Frame: 2 weeks per intervention, up to 7 weeks
Population: 5 completed participants
Measure: Mean (Standard Deviation); unit: percent time spent 70 mg/dL - 180 mg/dL
Groups:
- Overall Participants: Participants will follow specified diets for 2 weeks: standard carbohydrate, high protein/very low carbohydrate diet and high fat/very low carbohydrate diet.
Arm/Group | Overall Participants
Number analyzed (Participants) | 5
percent time spent 70 mg/dL - 180 mg/dL
  Baseline | 49.64 (19.92)
  Standard Carbohydrate Diet | 48.86 (15.41)
  High Protein Very Low Carbohydrate Diet | 60.78 (16.57)
  High Fat Very Low Carbohydrate Diet: number analyzed (Participants) | 4
  High Fat Very Low Carbohydrate Diet | 50.1 (16.83)

2. Secondary Outcome: Percentage of Time Spent > 180 mg/dL to 250 mg/dl
Description: The percent of time spent > 180 mg/dL to 250 mg/dl based on sensor-derived glucose values. Reflected is the percentage of time spent in the range of 181-250 mg/dL.
Time Frame: 2 weeks per intervention, up to 7 weeks
Population: 5 completed participants
Measure: Mean (Standard Deviation); unit: percent time spent > 180 to 250 mg/dL
Arm/Group | Overall Participants
Number analyzed (Participants) | 5
percent time spent > 180 to 250 mg/dL
  Baseline | 25.7 (3.19)
  Standard Carbohydrate | 25.36 (5.15)
  High Protein/Very Low Carbohydrate | 21.94 (5.75)
  High Fat/Very Low Carbohydrate: number analyzed (Participants) | 4
  High Fat/Very Low Carbohydrate | 21.32 (2.65)

3. Secondary Outcome: Percent Time Spent > 250 mg/dL Based on Sensor-derived Glucose Values
Description: The percent of time spent > 250 mg/dL based on sensor-derived glucose values. Presented is the percentage of time people spent in the range.
Time Frame: 2 weeks per intervention, up to 7 weeks
Population: 5 completed participants
Measure: Mean (Standard Deviation); unit: percent time spent > 250 mg/dL
Arm/Group | Overall Participants
Number analyzed (Participants) | 5
percent time spent > 250 mg/dL
  Baseline | 22.58 (19.24)
  Standard Carbohydrate | 21.36 (14.07)
  High Protein/Very Low Carbohydrate | 14.32 (13.17)
  High Fat/Very Low Carbohydrate: number analyzed (Participants) | 4
  High Fat/Very Low Carbohydrate | 24.95 (17.68)

4. Secondary Outcome: Percent of Time Spent > = 55 to < 70 mg/dL Based on Sensor-derived Glucose Values
Description: The percent of time spent > = 55 to < 70 mg/dL based on sensor-derived glucose values. Reflected is the percentage of time within range.
Time Frame: 2 weeks per intervention, up to 7 weeks
Population: 5 completed participants
Measure: Mean (Standard Deviation); unit: percent time spent > = 55 to < 70 mg/dL
Arm/Group | Overall Participants
Number analyzed (Participants) | 5
percent time spent > = 55 to < 70 mg/dL
  Baseline | 1.22 (1.61)
  Standard Carbohydrate | 2.96 (3.19)
  High Protein/Very Low Carbohydrate | 2.26 (1.93)
  High Fat/Very Low Carbohydrate: number analyzed (Participants) | 4
  High Fat/Very Low Carbohydrate | 2.65 (2.28)

5. Secondary Outcome: Percent Time Spent < 55 mg/dL Based on Sensor-derived Glucose Values
Description: The percent of time spent < 55 mg/dL based on sensor-derived glucose values during the timeframe. Presented is the percentage of overall time spent in the specified range.
Time Frame: 2 weeks per intervention, up to 7 weeks
Population: 5 completed participants
Measure: Mean (Standard Deviation); unit: percentage time spent < 55 mg/dL
Arm/Group | Overall Participants
Number analyzed (Participants) | 5
percentage time spent < 55 mg/dL
  Baseline | 0.68 (1.29)
  Standard Carbohydrate | 1.46 (2.23)
  High Protein/Very Low Carbohydrate | 0.68 (0.59)
  High Fat/Very Low Carbohydrate: number analyzed (Participants) | 4
  High Fat/Very Low Carbohydrate | 1.15 (1.06)

6. Secondary Outcome: Total Daily Insulin Dose
Description: The total daily insulin dose will be defined as the average total daily insulin dose will be calculated over 2 weeks. Values represent the mean units/kg/day for the 2 week period.
Time Frame: 2 weeks per intervention, up to 7 weeks
Population: 5 completed participants
Measure: Mean (Standard Deviation); unit: units/kg/day
Arm/Group | Overall Participants
Number analyzed (Participants) | 5
units/kg/day
  Baseline | 0.78 (0.09)
  Standard Carbohydrate | 0.82 (0.06)
  High Protein/Very Low Carbohydrate | 0.60 (0.08)
  High Fat/Very Low Carbohydrate: number analyzed (Participants) | 4
  High Fat/Very Low Carbohydrate | 0.69 (0.12)

7. Secondary Outcome: Average Sensor Glucose Level
Description: The average sensor glucose level recorded by the continuous glucose monitor over the 2 week dietary period in mg/dL.
Time Frame: 2 weeks per intervention, up to 7 weeks
Population: 5 completed participants
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Overall Participants
Number analyzed (Participants) | 5
mg/dL
  Baseline | 193 (44)
  Standard Carbohydrate | 186 (35)
  High Protein/Very Low Carbohydrate | 169 (30)
  High Fat/Very Low Carbohydrate: number analyzed (Participants) | 4
  High Fat/Very Low Carbohydrate | 193 (41)

ADVERSE EVENTS:
Time Frame: Up to 7 weeks total
Groups:
- Overall Participants: Presented are the overall group of participants regardless of level of the intervention. Adverse events were not systematically collected as part of the study.
Arm/Group | Overall Participants
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/84/NCT04082884/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/84/NCT04082884/ICF_001.pdf